CLINICAL TRIAL: NCT04746105
Title: A Study to Evaluate the Respiratory Safety of TS-142 in Patients with Obstructive Sleep Apnea Hypopnea.
Brief Title: A Clinical Pharmacology Study of TS-142 in Patients with Obstructive Sleep Apnea Hypopnea.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TS142-208
Record Dates: First submitted 2021-02-05; First posted 2021-02-09 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2021-11

CONDITIONS: Patients with Mild Obstructive Sleep Apnea Hypopnea
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TS-142 (Experimental): Period in which subjects received TS-142 10 mg or The night when subjects received TS-142
  Interventions: Drug: TS-142
- Placebo (Experimental): Period in which subjects received placebo or The night when subjects received matched placebo
  Interventions: Drug: Dose-matched Placebo to TS-142

INTERVENTIONS:
Drug: TS-142 — Subjects received single-dose of 10 mg of TS-142 (oral tablet)
  Arms: TS-142
Drug: Dose-matched Placebo to TS-142 — Subjects received single-dose matched placebo to TS-142 (oral tablet)
  Arms: Placebo

SUMMARY:
A study to evaluate the respiratory safety of TS-142 in patients with mild obstructive sleep apnea hypopnea.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male and female, age 20 years or older at the time of informed consent
* Patients who meet the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria for obstructive sleep apnea hypopnea
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

* Patients who meet the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria excepting obstructive sleep apnea hypopnea and insomnia disorder
* Patients who have clinically significant respiratory dysfunction (bronchiectasis, emphysema, asthma, etc.) other than obstructive sleep apnea hypopnea
* Patients with percutaneous arterial oxygen saturation (SpO2) <94% by pulse oximetry at visit 1
* Other protocol defined exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Least square mean difference of Apnea hypopnea index (AHI) from placebo | Day 1
  AHI is a number of apnea and hypopnea events per hour during sleep determined by polyso㎜ography (PSG).

SECONDARY OUTCOMES:
Least square mean difference of the mean SpO2 in total sleep time from placebo | Day 1
  The SpO2 will be simultaneously measured with PSG. The mean SpO2 during sleep determined by PSG will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Direcoter, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No